CLINICAL TRIAL: NCT02261857
Title: Personalized Three-Dimensionally Printed CPAP Masks for Obstructive Sleep Apnea Therapy in Children With Craniofacial Anomalies
Brief Title: 3D-Printed CPAP Masks for Children With Obstructive Sleep Apnea
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Glenn Green (Other)
Collaborators: American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other); University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Glenn Green, Sponsor-Investigator, University of Michigan
Organization: University of Michigan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00078727
Record Dates: First submitted 2014-09-29; First posted 2014-10-10 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Sleep Apnea, Obstructive; Craniofacial Abnormalities; Pediatric Disorder
Keywords: Obstructive Sleep Apnea; Craniofacial Abnormalities; Pediatrics; Computer-Aided Design; Continuous Positive Airway Pressure; Three-Dimensional Printing; Additive Manufacturing
MeSH Terms: conditions — Sleep Apnea, Obstructive; Craniofacial Abnormalities | interventions — Continuous Positive Airway Pressure; Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): Intervention: Subjects will undergo assessment and a personalized CPAP mask device will be manufactured using patient-specific computer-aided design and 3D printing. The subject will use the personalized CPAP mask for 1 month of consistent use and post-intervention data will be collected for compare to historical control (see other arm)
  Interventions: Device: Personalized continuous positive airway pressure (CPAP) mask
- Historical Control Arm (No Intervention): Pre-interventional baseline data on subject OSA, CPAP compliance, and quality of life (QoL) measures will be collected to serve as historical controls.

INTERVENTIONS:
Device: Personalized continuous positive airway pressure (CPAP) mask — Personalized CPAP mask manufactured for study subjects using a combination of patient-specific computer-aided design and three-dimensional printing
  Arms: Intervention Arm

SUMMARY:
The purpose of this study is to determine whether patient-specific computer-aided design (CAD) and three-dimensional (3D) printing can be utilized to produce personalized, effective continuous positive airway pressure (CPAP) masks for children with severe obstructive sleep apnea (OSA) and craniofacial anomalies who encounter significant difficulty using CPAP because of poorly fitting masks despite exhausting available commercial mask options.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common problem in the general pediatric population, generally cited as between 1-5%, with morbidity ranging from daytime behavioral problems and inattention to cardiopulmonary effects including hypertension and ventricular hypertrophy. OSA is dramatically more prevalent among children with certain craniofacial anomalies and syndromes (e.g. Pierre-Robin, Treacher Collins, etc.), generally because of small, short jaws, midface hypoplasia, and/or disproportionally large tongues . While tonsillectomy and adenoidectomy is considered first line therapy for OSA in the general pediatric population, children with OSA due to craniofacial anomalies frequently require more aggressive intervention to improve their breathing at night, which often includes continuous positive airway pressure ventilation (CPAP). Most children who require CPAP therapy are able to find a mask that will adequately seal while providing acceptable comfort, however a small percentage of children encounter significant difficulty finding a functional CPAP interface, most often because of dysmorphic facial features. This can prove a significant barrier to effective CPAP therapy and lead to frustration on the part of patients' caregivers and providers, as well as the associated morbidity of untreated severe OSA. The purpose of this feasibility study is to investigate the use of patient-specific computational design and three-dimensional (3D) printing to produce personalized CPAP masks for children intolerant of standard CPAP masks due to poor fit secondary to craniofacial anomalies who encounter significant difficulty using CPAP because of poorly fitting masks despite exhausting available commercial mask options.

Study Design

This will be a prospective case study examining the feasibility of using patient-specific CAD and 3D printing technology to produce personalized CPAP masks for children intolerant of commercially available masks due to poor fit. Patients will be recruited from the pediatric otolaryngology, pediatric oral maxillofacial surgery, and pediatric sleep clinics at the University of Michigan Medical Center, with a target cohort of five.

Only patients of study team members will be included in the study, and no recruitment will take place outside the clinics of participating study team members. We anticipate the study period to last 3 years, though it may terminate sooner if recruitment targets are reached expeditiously.

After recruitment and consent of a potential study subject, each subject will undergo an initial mask-design evaluation with members of the research team. At this initial visit, the following will be performed:

1. A head & neck physical exam, which a focus on characteristics important for treatment of OSA (e.g. jaw size and position, tongue size and position, characteristics of palate, presence or absence of cleft, external nasal deformity, external or internal nasal valvular collapse)
2. Review of patient's photographs
3. Generation of a topographic model of the patient's facial anatomy utilizing the 3dMDface system (specifics below) which will be export as a Stereolithography (.STL) file.

The patient's facial .STL file will then be imported into a computer-aided design (CAD) modeling program (MimicsTM or MagicsTM, Materialise, Belgium). Contact points along the topographic model are drawn out and utilized for modeling of the custom mask. The custom mask model is then exported in .STL format for import into the 3D printer for fabrication using a fused-deposition modeling (FDM) method (Object Pro, Stratasys, Israel).

Once the mask has been fabricated, patients will undergo a mask-fit evaluation. If a mask appears to fit well, the patient will use it at home with home CPAP for one month of consistent use. They will then return for debriefing and re-evaluation, with subsequent iterations of mask design as needed. If the mask functions for the patient better than any other alternatives, the patient will be allowed to continue to use the mask for up to one year, with ongoing surveillance by the research team, assessing for mask durability and ongoing usage/compliance.

Data collection will include:

* Objective data regarding the nature of each patient's obstructive sleep apnea and CPAP pressure requirements sleep-disordered breathing from the most recent available polysomnograms (sleep study, abbreviated PSG)
* Information regarding all prior CPAP masks attempted
* One month compliance data downloads from CPAP machines - with both the prior "best alternative" if usable, and with the customized mask, including percentage of days used, average hours usage, residual apnea-hypopnea index (AHI) and time spent in large leak per night.
* Standardized interview with patients and their parents regarding other masks used and experience with the customized mask(s).
* Descriptive anatomic information regarding facial anomalies contributing to poor mask fit, obtained from physical exam, photographs, and imaging studies.
* Validated quality of life measures taken before and at completion of trial period with customized CPAP mask, including the Pediatric Sleep Questionnaire (PSQ) and the OSA-18 , to assess the impact of successful CPAP use for our patients.

Analysis will involve basic descriptive statistics to describe both the objective outcomes (e.g. compliance data from CPAP machines) and quality of life measures (PSQ and OSA-18 surveys) as well as information on individual experiences collected during interviews.

Additional Data on 3D Photography System

Patient facial modeling information will be obtained utilizing a 3dMDface system (3dMD, Atlanta, GA). The 3dMD system is a three-dimensional photography system which generates a three-dimensional model of the patient's face utilizing multiple convergent cameras (see Figure 1 below). The three-dimensional model is generated utilizing hybrid stereophotogrammetry, with software algorithms using both projected random patterns and texture of the skin (pores, freckles, etc.) to stereo-triangulate and generate a 3D surface image. The 3D model of the patient's face is created within the 3dMDvultus software system, which can then export the model in .STL format. No patient identifying information is stored within the .STL file.

All 3D photography sessions with study subjects will be performed or supervised by one of the members of the study team. There will be no cost associated with using the 3dMDface system. Utilizing 3D photography allows us to obtain the most time-accurate topographic information of the patient's face while avoiding the cost and risk associated with conventional CT or MRI imaging.

Data Included in Registry:

* Pre- and post- intervention OSA-18 and PSQ questionnaire aggregates. Data to be recorded includes: sum score and mean score for each questionnaire.
* Pre-intervention AHI and oxygen saturation (SpO2) nadir based on most recent sleep PSG.
* Pre-intervention CPAP requirements based on most recent CPAP titration PSG.
* Pre-intervention compliance data downloads from subject's CPAP machines from prior 1 month's use. Data to be recorded includes: percentage of days used, average hours usage, residual apnea-hypopnea index (AHI), size of leak in liters per minute, and time spent in large leak per night.
* Post-intervention compliance data downloads from subject's CPAP machines from prior 1 month's use. Data to be recorded includes: percentage of days used, average hours usage, residual apnea-hypopnea index (AHI), size of leak in liters per minute, and time spent in large leak per night.

Data Registry QA:

• Physical and electronic PDF versions of each data registry primary source (questionnaires, polysomnograms, and CPAP compliance reports) will be kept for the 5 years past the duration of the study. Data uploaded to the patient registry will be verified with the institutional IRB.

ELIGIBILITY:
Inclusion Criteria:

* On-going need for CPAP therapy based on polysomnography
* Inability to tolerate CPAP attributed to poor fit by a sleep clinician
* The opinion of a sleep clinician that reasonable commercially available mask options have been exhausted
* Caregivers must also be proficient in English to complete standard questionnaires.

Exclusion Criteria:

* Subjects no longer needing CPAP therapy
* Subjects able to successfully use a commercially available mask.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in CPAP Compliance at 1 month | 1 month
  Subject CPAP usage data will be downloaded from their CPAP machine before beginning the use to personalized mask (baseline) and after 1 month of consistent use of the personalized mask (1 month post-intervention). Average hours usage will be recorded and compared between baseline CPAP usage data and 1 month post-intervention CPAP usage data to assess efficacy of the personalized mask compared to the best prior alternative. Outcome will be measured as a numerical value in hours per night.
Change in CPAP Leak Rate at 1 month | 1 month
  Subject CPAP usage data will be downloaded from their CPAP machine before beginning the use to personalized mask (baseline) and after 1 month of consistent use of the personalized mask (1 month post-intervention). Leak in liters per minute will be recorded and compared between baseline CPAP usage data and 1 month post-intervention CPAP usage data to assess efficacy of the personalized mask compared to the best prior alternative. Outcome will be measured as a numerical value in liters per minute.
Change in residual AHI on CPAP at 1 month | 1 month
  Subject CPAP usage data will be downloaded from their CPAP machine before beginning the use to personalized mask (baseline) and after 1 month of consistent use of the personalized mask (1 month post-intervention). Residual apnea-hypopnea index (AHI) will be recorded and compared between baseline CPAP usage data and 1 month post-intervention CPAP usage data to assess efficacy of the personalized mask compared to the best prior alternative. Outcome will be measured as a numerical value denoting AHI.
Change in time spent in large leak on CPAP at 1 month | 1 month
  Subject CPAP usage data will be downloaded from their CPAP machine before beginning the use to personalized mask (baseline) and after 1 month of consistent use of the personalized mask (1 month post-intervention). Percentage (%) time spent in large leak per night will be recorded and compared between baseline CPAP usage data and 1 month post-intervention CPAP usage data to assess efficacy of the personalized mask compared to the best prior alternative. Outcome will be measured as a numerical percentage as a percentage of total time spent in large leak per night over total time using CPAP per night.

SECONDARY OUTCOMES:
Change in Quality of Life via OSA-18 questionnaire | 1 month
  Subject's parents or legal guardians will complete OSA-18 questionnaire (validated OSA quality of of life questionnaires) pre-intervention (baseline) and at 1-month post-intervention. These will be compared to assess effect on quality of life of the interventional device. Outcome will be measured as a numerical value as sum of all question value responses.
Safety outcomes: Comfort at baseline | Baseline
  Subjects will be assessed clinically when first wearing the interventional device to ensure there are no issues with device fit, comfort, or undue forces on the face. Outcome will be measured as a binary numerical value with 0 denoting no issues with comfort and 1 denoting issues with comfort.
Safety outcomes: Comfort at 1 month | 1 month
  Subjects will be assessed clinically after using the personalized mask consistently for 1 month at home to ensure there are no issues with device fit, comfort or undue forces on the face. Subject's parents or legal guardians are instructed to contact the study team for earlier follow-up at anytime if any concerns about device fit or use occur. Outcome will be measured as a binary numerical value with 0 denoting no issues with comfort and 1 denoting issues with comfort.
Safety outcomes: Skin reaction at 1 month | 1 month
  Subjects will be assessed clinically after using the personalized mask consistently for 1 month at home to ensure there are no issues with skin reaction or breakdown on the face. Subject's parents or legal guardians are instructed to contact the study team for earlier follow-up at anytime if any concerns about device fit or use occur. Outcome will be measured as a binary numerical value with 0 denoting no issues with skin reaction and 1 denoting issues with skin reaction.
Change in Quality of Life via PSQ questionnaire | 1 month
  Subject's parents or legal guardians will complete PSQ questionnaire (validated OSA quality of of life questionnaires) pre-intervention (baseline) and at 1-month post-intervention. These will be compared to assess effect on quality of life of the interventional device. Outcome will be measured as a numerical value as sum of all question value responses.
Safety outcomes: durability at 1 month | 1 month
  Subjects will be assessed clinically after using the personalized mask consistently for 1 month at home to ensure there are no issues with excessive wear or tear of the personalized mask. Subject's parents or legal guardians are instructed to contact the study team for earlier follow-up at anytime if any concerns about device fit or use occur. Outcome will be measured as a binary numerical value with 0 denoting no issues with durability and 1 denoting issues with durability.
Safety outcomes: Skin reaction at 12 months | 12 months
  Subjects will be assessed clinically after using the personalized mask consistently for 12 months at home to ensure there are no issues with skin reaction or breakdown on the face. Subject's parents or legal guardians are instructed to contact the study team for earlier follow-up at anytime if any concerns about device fit or use occur. Outcome will be measured as a binary numerical value with 0 denoting no issues with skin reaction and 1 denoting issues with skin reaction.
Safety outcomes: Durability at 12 months | 12 months
  Subjects will be assessed clinically after using the personalized mask consistently for 12 months at home to ensure there are no issues with excessive wear or tear of the personalized mask. Subject's parents or legal guardians are instructed to contact the study team for earlier follow-up at anytime if any concerns about device fit or use occur. Outcome will be measured as a binary numerical value with 0 denoting no issues with durability and 1 denoting issues with durability.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn E Green, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Ward SD, Sheldon SH, Shiffman RN, Lehmann C, Spruyt K; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):e714-55. doi: 10.1542/peds.2012-1672. Epub 2012 Aug 27. PMID 22926176
- [Background] Brunetti L, Rana S, Lospalluti ML, Pietrafesa A, Francavilla R, Fanelli M, Armenio L. Prevalence of obstructive sleep apnea syndrome in a cohort of 1,207 children of southern Italy. Chest. 2001 Dec;120(6):1930-5. doi: 10.1378/chest.120.6.1930. PMID 11742924
- [Background] Amin RS, Kimball TR, Bean JA, Jeffries JL, Willging JP, Cotton RT, Witt SA, Glascock BJ, Daniels SR. Left ventricular hypertrophy and abnormal ventricular geometry in children and adolescents with obstructive sleep apnea. Am J Respir Crit Care Med. 2002 May 15;165(10):1395-9. doi: 10.1164/rccm.2105118. PMID 12016102
- [Background] Duman D, Naiboglu B, Esen HS, Toros SZ, Demirtunc R. Impaired right ventricular function in adenotonsillar hypertrophy. Int J Cardiovasc Imaging. 2008 Mar;24(3):261-7. doi: 10.1007/s10554-007-9265-1. Epub 2007 Sep 6. PMID 17846918
- [Background] Leung LC, Ng DK, Lau MW, Chan CH, Kwok KL, Chow PY, Cheung JM. Twenty-four-hour ambulatory BP in snoring children with obstructive sleep apnea syndrome. Chest. 2006 Oct;130(4):1009-17. doi: 10.1378/chest.130.4.1009. PMID 17035432
- [Background] Luna-Paredes C, Anton-Pacheco JL, Garcia Hernandez G, Martinez Gimeno A, Romance Garcia AI, Garcia Recuero II. Screening for symptoms of obstructive sleep apnea in children with severe craniofacial anomalies: assessment in a multidisciplinary unit. Int J Pediatr Otorhinolaryngol. 2012 Dec;76(12):1767-70. doi: 10.1016/j.ijporl.2012.08.020. Epub 2012 Sep 11. PMID 22980525
- [Background] Plomp RG, Bredero-Boelhouwer HH, Joosten KF, Wolvius EB, Hoeve HL, Poublon RM, Mathijssen IM. Obstructive sleep apnoea in Treacher Collins syndrome: prevalence, severity and cause. Int J Oral Maxillofac Surg. 2012 Jun;41(6):696-701. doi: 10.1016/j.ijom.2012.01.018. Epub 2012 Apr 20. PMID 22521672
- [Background] Zandieh SO, Padwa BL, Katz ES. Adenotonsillectomy for obstructive sleep apnea in children with syndromic craniosynostosis. Plast Reconstr Surg. 2013 Apr;131(4):847-852. doi: 10.1097/PRS.0b013e3182818f3a. PMID 23542256
- [Background] Chervin RD, Hedger K, Dillon JE, Pituch KJ. Pediatric sleep questionnaire (PSQ): validity and reliability of scales for sleep-disordered breathing, snoring, sleepiness, and behavioral problems. Sleep Med. 2000 Feb 1;1(1):21-32. doi: 10.1016/s1389-9457(99)00009-x. PMID 10733617
- [Background] Franco RA Jr, Rosenfeld RM, Rao M. First place--resident clinical science award 1999. Quality of life for children with obstructive sleep apnea. Otolaryngol Head Neck Surg. 2000 Jul;123(1 Pt 1):9-16. doi: 10.1067/mhn.2000.105254. PMID 10889473